CLINICAL TRIAL: NCT06419075
Title: Local Infiltration of TranExamic Acid in Surgical Management of Pelvic Organ Prolapse: a Pilot Randomized Clinical Trial
Brief Title: Tranexamic Acid in Vaginal Reconstructive Surgery
Acronym: TEXAS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: closed study due to lack of faculty
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-0273
Record Dates: First submitted 2024-05-08; First posted 2024-05-17 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Pelvic Organ Prolapse
Keywords: Tranexamic Acid; Colpocleisis
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Tranexamic Acid; Vasopressins; Arginine Vasopressin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The enrolled subjects will be randomized into one of the 3 arms including tranexamic acid (2 mg/dL), vasopressin (0.1 U/dL), and normal saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The attending anesthesiologist will receive the randomized assignment from the lead research team at UTMB and prepare the diluted study agents. The OR staff, attending surgeon, and learners including fellows and residents are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal Saline (NaCl 0.9%) (Placebo Comparator): Local infiltration of 50 cc NaCl 0.9% into the vaginal submucosa during colpocleisis dissection
  Interventions: Other: NaCl 0.9%
- Tranexamic Acid (2 mg/dL) (Experimental): Local infiltration of 50 cc Tranexamic Acid (2 mg/dL) into the vaginal submucosa during colpocleisis dissection
  Interventions: Drug: Tranexamic acid
- Vasopressin (0.1 U/dL) (Experimental): Local infiltration of 50 cc Vasopressin (0.1 U/dL) into the vaginal submucosa during colpocleisis dissection
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Tranexamic acid — The intervention of 50 cc TXA (2 mg/mL) local infiltration is determined after carefully reviewing the literature. Scarafoni et al. recommends that the local TXA should not exceed at a concentration of 5-10 mg/mL to avoid cytotoxicity that may affect the wound re-epithelialization (22). In a prospective study on facelift bleeding, Kochuba et al. demonstrates that local TXA (1-2 mg/mL) with total 100 mg and 200 mg TXA safely and effectively decreased bleeding, operating room time, and drain output compared with traditional local anesthetic technique (14). Fathimani et all reports the local use of modified tumescent anesthesia solution with low TXA concentration (2 mg/dL) and total average dosage of TXA ranging 120-1000 mg is safe and promising in achieving less ecchymosis, edema, and seroma in common facial cosmetic surgical procedures (31). With a total dosage of 100 mg TXA and a volume of 50 cc injection, the concentration is calculated to be 2 mg/dL.
  Other Names: Tranexamic acid (CYKLOKAPRON) (Pfizer, New York, NY).
  Arms: Tranexamic Acid (2 mg/dL)
Drug: Vasopressin — The intervention of 50 cc Vasopressin (0.1U/mL) local infiltration is determined from several systematic reviews. Hafidh et al. shows that injection of diluted Vasopressin (3.6 to 10 units) with various concentration during hysterectomy significantly reduces the intraoperative blood loss when compared to placebo, and without increasing the hazard of cardiovascular toxicities. Cui et al. reports similar results, but including other vaginal surgeries. The common preparation for dilute Vasopressin is 0.1 U/mL or 1.0 U/mL from a 1cc vial of 20 U/mL Vasopressin. The advantage of 0.1 U/mL concentration is to avoid a relatively large bolus of concentrated 1.0 U/mL Vasopressin injected intravascularly by accident. A cumulative total dose of 4 to 6 units of Vasopressin administered in a dilute solution is proposed to be an upper limit. Therefore, the cumulative total dose of 5 units Vasopressin from 50 cc (0.1U/mL) is in the safe therapeutic range.
  Other Names: Vasopressin (Vasostrict) (Par Pharmaceutical, Chestnut Ridge, NY).
  Arms: Vasopressin (0.1 U/dL)
Other: NaCl 0.9% — The intervention of 50 cc NaCl 0.9% local infiltration serves a placebo control.
  Arms: Normal Saline (NaCl 0.9%)

SUMMARY:
Tranexamic acid (TXA) has been demonstrated to reduce blood loss in trauma, orthopedic, cardiac, and plastic surgeries in numerous well-designed and adequately powered studies. As a result of this evidence for benefit, TXA is routinely used to reduce blood loss during these surgeries. There are no studies regarding the use of TXA in urogynecology. The investigators seek to explore the effect and safety of local infiltration of TXA in vaginal reconstructive surgery.

DETAILED DESCRIPTION:
This is a multicenter, double blinded, pilot randomized clinical trial that will be conducted at UTMB Health, and other participating sites. Each participating site will obtain IRB approval. Women with symptomatic, stage II to IV Pelvic organ prolapse (POP) who plan colpocleisis will be approached to participate. Using the study protocol inclusion and exclusion criteria, patient's eligibility will be determined. All eligible subjects will provide the written informed consent before any research data is collected. All screening assessment will be completed at a preoperative, in-person, clinic visit, and within 60 days of surgery. The subject will then undergo randomization to the local TXA, or Vasopressin, or NS group with the total sample size of 36 female subjects (12 per group). Concomitant procedures for POP or urinary incontinence are permitted and will be based upon the operating surgeons' standard clinical practice and best clinical judgement. The anesthesia team is responsible for preparing the study agents, monitoring intraoperative cardiovascular parameters (blood pressure and heart rate) as well as adverse events, and determining the blood transfusion if needed. Subsequently, the subject will have postoperative follow up at 2 weeks and 6 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Females who are menopausal at the time of consent
2. Able to understand and read English
3. Able and willing to provide written informed consent
4. Able to comply with the follow-up study protocol, per clinician judgment
5. Symptomatic POP (bulge or pressure) evidenced with vaginal prolapse with POP-Q measurement consistent with Stage II-IV
6. LeFort or complete colpocleisis as desired surgical approach to correct POP with and without other concomitant procedures
7. History of abdominal or vaginal surgery for POP
8. American Society of Anesthesiologists (ASA) physical status I or II

Exclusion Criteria:

1. Texas Department of Criminal Justice prisoners
2. Refusal of blood products (e.g, Jehovah's witnesses)
3. ASA physical status III or IV
4. Known allergy or hypersensitivity to TXA or any of the ingredients
5. Subarachnoid hemorrhage
6. Active intravascular clotting, thromboembolic disease (cerebral thrombosis, deep vein thrombosis, or pulmonary embolism)
7. Epilepsy, seizure disorders requiring anti-epileptic medication(s)
8. Acquired impaired color vision (color blindness, retinal involvement)
9. Intrinsic risk of thrombosis or thromboembolism (hypercoagulopathy, thrombogenic cardiac rhythm disease, thrombogenic valvular disease)
10. History of severe liver disease
11. Known allergy or hypersensitivity to 8-L-arginine vasopressin or chlorobutanol
12. History of cardiac diseases (decompensated congestive heart failure CHF, recent coronary artery disease CAD within 30 days, recent myocardial infarction MI within 30 days)
13. History of reversible nephrogenic diabetes insipidus
14. History of primary pelvic organ cancer (uterine, ovarian, endometrial, cervical, bladder) or any cancer that is metastatic to the pelvis
15. Prior or current pelvic radiation, or chemotherapy.
16. Females who desires to have vaginal sexual intercourse after the surgery

Ages: 50 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Intraoperative quantitative blood loss QBL (mL) | Intraoperatively
  Compare intraoperative QBL during colpocleisis with the local infiltration of Tranexamic acid to the current standard of care, vasopressin or normal saline.

SECONDARY OUTCOMES:
Colpocleisis operative time (min) | Intraoperatively
  Compare the colpocleisis operative time between Tranexamic acid, vasopressin or normal saline groups
Intraoperative blood pressure (mmHg) | Intraoperatively
  Evaluate the effect blood pressures at 1, 5, and 10 mins after the local infiltration of Tranexamic acid, vasopressin and NS into the vaginal mucosa.
Intraoperative hear rate (beats/min) | Intraoperatively
  Evaluate the effect on heart rate at 1, 5, and 10 mins after the local infiltration of Tranexamic acid, vasopressin and NS into the vaginal mucosa.
Postoperative complications | 2 weeks and 6 weeks postoperatively
  Assess postoperative complications following colpocleisis using the Clavien-Dindo Classification (CDC) categories
Rate of transfusion | Intraoperatively and 2 weeks postoperatively
  Quantify the need for blood-product transfusion and the volume administered as a direct result of colpocleisis, either intraoperative or postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Kilic, MD, Principal Investigator — University of Texas Medical Branch Galveston; Ann Tran, MD, Principal Investigator — Mount Sinai Hospital & Medical Center

IPD SHARING:
Plan to Share IPD: No
We are not planning to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Smith FJ, Holman CD, Moorin RE, Tsokos N. Lifetime risk of undergoing surgery for pelvic organ prolapse. Obstet Gynecol. 2010 Nov;116(5):1096-100. doi: 10.1097/AOG.0b013e3181f73729. PMID 20966694
- [Background] Cheng W, Bu C, Hong F, Zhong X, Jin C, Yang X, Sun X, Wang J. Perioperative hemorrhagic complications in pelvic floor reconstructive surgery. Int Urogynecol J. 2019 Jul;30(7):1141-1146. doi: 10.1007/s00192-018-3667-6. Epub 2018 May 21. PMID 29785542
- [Background] Lambrou NC, Buller JL, Thompson JR, Cundiff GW, Chou B, Montz FJ. Prevalence of perioperative complications among women undergoing reconstructive pelvic surgery. Am J Obstet Gynecol. 2000 Dec;183(6):1355-8; discussion 1359-60. doi: 10.1067/mob.2000.110911. PMID 11120496
- [Background] Johnson DJ, Scott AV, Barodka VM, Park S, Wasey JO, Ness PM, Gniadek T, Frank SM. Morbidity and Mortality after High-dose Transfusion. Anesthesiology. 2016 Feb;124(2):387-95. doi: 10.1097/ALN.0000000000000945. PMID 26569167
- [Background] Ghadimi K, Levy JH, Welsby IJ. Perioperative management of the bleeding patient. Br J Anaesth. 2016 Dec;117(suppl 3):iii18-iii30. doi: 10.1093/bja/aew358. PMID 27940453
- [Background] Cui Y, Chen I, Chernoff A, Clancy A. Effectiveness of prophylactic pharmacological hemostatic agents for reduction of blood loss at vaginal surgery: a systematic review and meta-analysis. Int Urogynecol J. 2023 Dec;34(12):2945-2957. doi: 10.1007/s00192-023-05614-1. Epub 2023 Aug 16. PMID 37584705
- [Background] Hafidh B, Latifah HM, Gari A, Alshahrani MS, AlSghan R, Alkhamis WH, Allam HS, AlRasheed MA, Bakhsh H, Abu-Zaid A, Baradwan S. Vasopressin to Control Blood Loss during Hysterectomy: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Minim Invasive Gynecol. 2022 Mar;29(3):355-364.e2. doi: 10.1016/j.jmig.2021.10.003. Epub 2021 Oct 12. PMID 34648933
- [Background] Willis-Gray MG, Husk KE, Brueseke TJ, Connolly A, Geller EJ. Lidocaine Use in Vaginal Surgery and Risk of Toxicity. Female Pelvic Med Reconstr Surg. 2020 Sep;26(9):546-549. doi: 10.1097/SPV.0000000000000622. PMID 30346319
- [Background] Zakhari A, Sanders AP, Solnik MJ. Tranexamic acid in gynecologic surgery. Curr Med Res Opin. 2020 Mar;36(3):513-520. doi: 10.1080/03007995.2019.1708533. Epub 2020 Jan 6. PMID 31865770
- [Background] Luetzenberg FS, Lyford-Pike S. Modern use of tranexamic acid in facial plastic surgery. Curr Opin Otolaryngol Head Neck Surg. 2023 Aug 1;31(4):219-223. doi: 10.1097/MOO.0000000000000886. Epub 2023 Apr 13. PMID 37052603
- [Background] Breau RH, Kokolo MB, Punjani N, Cagiannos I, Beck A, Niznick N, Buenaventura C, Cowan J, Knoll G, Momoli F, Morash C, Ruzicka M, Schachkina S, Tinmouth A, Xie HY, Fergusson DA. The effects of lysine analogs during pelvic surgery: a systematic review and meta-analysis. Transfus Med Rev. 2014 Jul;28(3):145-55. doi: 10.1016/j.tmrv.2014.05.002. Epub 2014 May 18. PMID 24958068
- [Background] El Minawi HM, Kadry HM, El-Essawy NM, El Saadany ZA, Nouh OM. The effect of tranexamic acid on blood loss in liposuction: a randomized controlled study. Eur J Plast Surg. 2023;46(2):227-237. doi: 10.1007/s00238-022-01995-6. Epub 2022 Oct 22. PMID 36311870
- [Background] Couto RA, Charafeddine A, Sinclair NR, Nayak LM, Zins JE. Local Infiltration of Tranexamic Acid With Local Anesthetic Reduces Intraoperative Facelift Bleeding: A Preliminary Report. Aesthet Surg J. 2020 May 16;40(6):587-593. doi: 10.1093/asj/sjz232. PMID 31504134
- [Background] Kochuba AL, Coombs DM, Kwiecien GJ, Sinclair NR, Zins JE. Prospective Study Assessing the Effect of Local Infiltration of Tranexamic Acid on Facelift Bleeding. Aesthet Surg J. 2021 Mar 12;41(4):391-397. doi: 10.1093/asj/sjaa198. PMID 32644111
- [Background] Coombs DM, Kwiecien GJ, Sinclair NR, Jin A, Zins JE. Local Infiltration of Tranexamic Acid During Facelift Improves Operating Room Efficiency: A Matched Patient Study. Aesthet Surg J. 2022 Aug 24;42(9):971-977. doi: 10.1093/asj/sjac067. PMID 35350068
- [Background] Ausen K, Fossmark R, Spigset O, Pleym H. Safety and Efficacy of Local Tranexamic Acid for the Prevention of Surgical Bleeding in Soft-Tissue Surgery: A Review of the Literature and Recommendations for Plastic Surgery. Plast Reconstr Surg. 2022 Mar 1;149(3):774-787. doi: 10.1097/PRS.0000000000008884. PMID 35196701
- [Background] Rohrich RJ, Cho MJ. The Role of Tranexamic Acid in Plastic Surgery: Review and Technical Considerations. Plast Reconstr Surg. 2018 Feb;141(2):507-515. doi: 10.1097/PRS.0000000000003926. PMID 28938364
- [Background] Buchsbaum GM, Lee TG. Vaginal Obliterative Procedures for Pelvic Organ Prolapse: A Systematic Review. Obstet Gynecol Surv. 2017 Mar;72(3):175-183. doi: 10.1097/OGX.0000000000000406. PMID 28304415
- [Background] Grzybowska ME, Futyma K, Kusiak A, Wydra DG. Colpocleisis as an obliterative surgery for pelvic organ prolapse: is it still a viable option in the twenty-first century? Narrative review. Int Urogynecol J. 2022 Jan;33(1):31-46. doi: 10.1007/s00192-021-04907-7. Epub 2021 Aug 18. PMID 34406418
- [Background] von Pechmann WS, Mutone M, Fyffe J, Hale DS. Total colpocleisis with high levator plication for the treatment of advanced pelvic organ prolapse. Am J Obstet Gynecol. 2003 Jul;189(1):121-6. doi: 10.1067/mob.2003.546. PMID 12861149
- [Background] Hill AJ, Walters MD, Unger CA. Perioperative adverse events associated with colpocleisis for uterovaginal and posthysterectomy vaginal vault prolapse. Am J Obstet Gynecol. 2016 Apr;214(4):501.e1-501.e6. doi: 10.1016/j.ajog.2015.10.921. Epub 2015 Oct 31. PMID 26529371
- [Background] Elena Scarafoni E. A Systematic Review of Tranexamic Acid in Plastic Surgery: What's New? Plast Reconstr Surg Glob Open. 2021 Mar 23;9(3):e3172. doi: 10.1097/GOX.0000000000003172. eCollection 2021 Mar. PMID 33907653
- [Background] Frishman G. Vasopressin: if some is good, is more better? Obstet Gynecol. 2009 Feb;113(2 Pt 2):476-477. doi: 10.1097/AOG.0b013e31819698bb. No abstract available. PMID 19155925
- [Background] Quantitative Blood Loss in Obstetric Hemorrhage: ACOG COMMITTEE OPINION, Number 794. Obstet Gynecol. 2019 Dec;134(6):e150-e156. doi: 10.1097/AOG.0000000000003564. PMID 31764759
- [Background] Ker K, Beecher D, Roberts I. Topical application of tranexamic acid for the reduction of bleeding. Cochrane Database Syst Rev. 2013 Jul 23;2013(7):CD010562. doi: 10.1002/14651858.CD010562.pub2. PMID 23881695
- [Background] DILLON TF, MARBURY BE, BONSNES RW, DOUGLAS RG, DU VIGNEAUD V. Vasopressin as a hemostatic in gynecologic surgery; a preliminary report. Obstet Gynecol. 1958 Apr;11(4):363-71. No abstract available. PMID 13517741